CLINICAL TRIAL: NCT00748020
Title: Narrow-Band UVB-Therapy in Psoriasis: Randomised Double-Blind Comparison of Erythematogenic and Suberythematogenic Irradiation Regimens
Brief Title: Narrow-Band UVB-Therapy in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: M.J.P. Gerritsen, MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UVB-MKL
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group 1 (Active Comparator): Erythematogenic irradiation scheme
  Interventions: Procedure: UVB phototherapy
- group 2 (Active Comparator): Suberythematogenic irradiation scheme
  Interventions: Procedure: UVB phototherapy

INTERVENTIONS:
Procedure: UVB phototherapy — Group 1: every irradiation an increase of 40%, starting with 70% of the minimal erythema dose
  Arms: group 1
Procedure: UVB phototherapy — Group 2: every irradiation an increase of 20%, starting with 30% of the minimal erythema dose
  Arms: group 2

SUMMARY:
Study on two different irradiation schemes in UVB phototherapy for psoriasis. Previous studies demonstrated a similar clinical effect in erythematogenic and suberythematogenic irradiation, with less complications in suberythematogenic irradiation. Most of these studies used both irradiation schemes within the same patient. UVB has a systemic effect on the body. Our hypothesis is that previous conclusions are incorrect and that the erythematogenic scheme will result in earlier clearance of the psoriasis.

DETAILED DESCRIPTION:
109 psoriasis patients, referred for UVB phototherapy, participated in our study after given their written informed consent. After determining the minimal erythema dose (MED) patients were randomised in either group 1, erythematogenic scheme, or group 2, suberythematogenic scheme. Group 1 started with 70% of MED and every following irradiation with an increase of 40%. Group 2 started with 30% of MED and every next visit an increase of 20%. The study protocol was adjusted in case of erythema (sunburn) according to a standard erythema-phototherapy protocol, varying from skip one irradiation to lowering the percentage of increase. In case of clearance the study stopped. Clearance was defined as less than 10% of baseline body area of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for UVB phototherapy
* Older than 18 years

Exclusion Criteria:

* No topical medication for 2 weeks
* No systemic medication for 4 weeks
* No medication (betablocker, lithium) interfering with psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2003-01; Primary Completion 2006-05 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
clearance is defined as less than 10% affected body area with psoriasis compared with baseline | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rianne Gerritsen, MD, PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Department of Dermatology, Nijmegen, Nijmegen, Netherlands